CLINICAL TRIAL: NCT00854295
Title: Prospective Multicenter Post Approval Study of the LPS-Flex Mobile Bearing Knee
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-100
Record Dates: First submitted 2009-02-26; First posted 2009-03-03 (Estimated); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Osteoarthritis; Traumatic Arthritis; Avascular Necrosis of the Femoral Condyle; Moderate Varus; Valgus; Flexion Deformities
Keywords: arthritis; osteoarthritis; degenerative knee disease; avascular necrosis; total knee replacement; TKA
MeSH Terms: conditions — Osteoarthritis; Genu Valgum; Arthritis; Osteonecrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

ARMS (2):
- Post-Approval Study Group (Group 2) (Experimental): Subjects enrolled in a short-term study (5 years) consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by orthopedic surgeons experienced in primary total knee replacement. All Group 2 subjects, both unilateral and bilateral subjects, are in the same arm of the study. As part of the PAS study, these subjects were followed from Pre-operative to 5 years.
  Interventions: Device: NexGen LPS-Flex Mobile Bearing Knee
- Investigational Device Exemption Group (Group 1) (Experimental): Subjects who were implanted with either the LPS Flex Fixed Bearing Knee (control population) or the LPS Flex Mobile Bearing Knee device during the previous Investigational Device Exemption study. As part of the PAS study, these subjects were followed from 4 years to 10 years.
  Interventions: Device: NexGen LPS-Flex Mobile Bearing Knee

INTERVENTIONS:
Device: NexGen LPS-Flex Mobile Bearing Knee — Total Knee Replacement
  Other Names: Mobile bearing knee

SUMMARY:
The purpose of the study is to assess the long-term performance of the NexGen LPS-Flex Mobile Bearing Knee in the treatment of patients with severe knee pain or degenerative knee disease.

DETAILED DESCRIPTION:
The NexGen LPS-FLex Mobile Bearing Knee received FDA approval for commercial distribution in the US on December 10, 2007. The approval was in accordance with a "condition of approval" to perform a 10-year post approval study to evaluate the longer-term safety and effectiveness of the LPS-Flex Mobile Bearing Knee. The post approval study will consist of patients from the investigational device exemption study arm (Group 1) as well as patients who are eligible for a total knee replacement and have been chosen to receive the LPS-Flex Mobile Knee (Group 2). Group 1 will be followed from 4 years through a total of 10 years from the date of surgery. Group 2 will be followed from pre-op through a total of 5 years from the date of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritis
* Primary and secondary traumatic arthritis
* Avascular necrosis of the femoral condyle
* Moderate varus, valgus, or flexion deformities (i.e. valgus/varus deformity of less than or equal to 15 degrees, fixed flexion deformity of less than or equal to 10 degrees)

Exclusion Criteria:

* Previous history of infection in the affected joint and/or local/systemic infection that may affect the prosthetic joint
* Insufficient bone stock on femoral or tibial surfaces
* Skeletal immaturity
* Neuropathic arthropathy
* Osteoporosis or any loss of musculature or neuromuscular disease that compromises the affected limb
* A stable, painless arthrodesis in a satisfactory functional position
* Severe instability secondary to the absence of collateral integrity
* Total knee arthroplasty is contraindicated in patients who have rheumatoid arthritis (RA) and an ulcer of the skin or a history of recurrent breakdown of the skin because their risk of postoperative infection is greater. RA patient using steroids may also have increased risk of infection. Late infections in RA patients have been reported 24+ months postoperative.
* Patient is a poor compliance risk, i.e., history of ethanol or drug abuse, or mental handicap that would compromise patient compliance with respect to rehabilitation or follow-up
* Patient is not willing or able to give informed consent to participate in the follow-up program
* Patient is not willing to return for all scheduled follow-up appointments as defined by this protocol.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 266 (Actual)
Dates: Start 2009-04 (Actual); Primary Completion 2020-06 (Actual); Study Completion 2021-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (3):
- United States (3):
  - Phoenix Clinical Research, Tamarac, Florida
  - Advanced Orthopaedics, Auburn Hills, Michigan
  - Tennessee Orthopaedic Foundation for Education and Research, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeons experienced in primary total knee replacement. Subjects who had one operative knee were in the Unilateral Group and subjects who had two operative knees were in the Bilateral Group. These subjects are considered "Group 2" per the study protocol.
Pre-assignment Details: All cases in "Group 1" per the protocol (subjects in the previous IDE study who were eligible to participate in the PAS) have study completed and are not included in these results. A final report for Group 1 was previously approved by FDA on June 29, 2016. Since 2016, only data from Group 2 subjects (PAS Group) was reported to FDA and are applicable to this clinicatrials.gov record.
Groups:
- LPS Flex Mobile Unilateral Group (Group 2): Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee.
- LPS Flex Mobile Bilateral Group (Group 2): Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in both knees.
- LPS Flex Fixed (Group 1): Subjects in this group received the LPS-Flex Fixed Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee and were enrolled in a previous Investigational Device Exemption study.
- LPS Flex Mobile (Group 1): Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee and were enrolled in a previous Investigational Device Exemption study.
Period: Overall Study
Arm/Group | LPS Flex Mobile Unilateral Group (Group 2) | LPS Flex Mobile Bilateral Group (Group 2) | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
Started | 106 | 14 | 77 | 69
Completed | 65 | 8 | 54 | 44
Not Completed | 41 | 6 | 23 | 25
Not completed — Death | 7 | 0 | 1 | 1
Not completed — Adverse Event | 6 | 1 | 1 | 3
Not completed — Lost to Follow-up | 18 | 5 | 21 | 21
Not completed — Physician Decision | 10 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement.
Groups:
- LPS Flex Mobile Uniliteral (Group 2): Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement. Subjects who were implanted with the study device in one knee were in the Unilateral Group.
- LPS Flex Mobile Bilateral (Group 2): Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement. Subjects who were implanted with the study device in two knees were in the Bilateral Group.
- Total: Total of all reporting groups
Arm/Group | LPS Flex Mobile Uniliteral (Group 2) | LPS Flex Mobile Bilateral (Group 2) | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1) | Total
Number analyzed (Participants) | 106 | 14 | 77 | 69 | 266
Age, Continuous [Mean (Full Range); unit: Years] | 65.8 [45 to 85] | 62.4 [52 to 72] | 61.4 [35 to 81] | 62.5 [34 to 80] | 65.4 [45 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68 | 12 | 51 | 40 | 171
  Male | 38 | 2 | 26 | 29 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 12 | 0 | 5 | 1 | 18
  White | 91 | 12 | 70 | 66 | 239
  More than one race | 2 | 2 | 1 | 2 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 106 | 14 | 77 | 69 | 266

OUTCOME MEASURES:

1. Primary Outcome: Group 2 - Total Knee Society Score (KSS)
Description: Total Knee Society Score is used to assess pain and function which is scored from 0 to 200 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions.
Time Frame: Pre-op, 6 week, 6 month, 1 year, 2 year, 3 year, 4 year, and 5 year
Population: Only subjects with an evaluable endpoint at each time frame interval were used to calculate mean and standard deviations.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- LPS Flex Mobile Unilateral Group (Group 2): Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement. Subjects who were implanted with the study device in one knee were in the Unilateral Group.
- LPS Flex Mobile Bilateral Group (Group 2): Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement. Subjects who were implanted with the study device in two knees were in the Bilateral Group.
Arm/Group | LPS Flex Mobile Unilateral Group (Group 2) | LPS Flex Mobile Bilateral Group (Group 2)
Number analyzed (Participants) | 106 | 14
score on a scale
  Pre-op | 92.2 (28.5) | 78.5 (29)
  6 Week: number analyzed (Participants) | 100 | 13
  6 Week | 118.2 (33) | 96.7 (34)
  6 Month: number analyzed (Participants) | 98 | 10
  6 Month | 148 (29.7) | 130.4 (51.5)
  1 Year: number analyzed (Participants) | 96 | 10
  1 Year | 159.2 (28.1) | 137.2 (56.9)
  2 Year: number analyzed (Participants) | 85 | 11
  2 Year | 159.2 (32.2) | 149.4 (34.7)
  3 Year: number analyzed (Participants) | 80 | 10
  3 Year | 161.1 (27.3) | 147.3 (45.3)
  4 Year: number analyzed (Participants) | 72 | 10
  4 Year | 160.2 (29.4) | 121.3 (56.7)
  5 Year: number analyzed (Participants) | 65 | 8
  5 Year | 160.8 (28.6) | 167.1 (29.3)

2. Primary Outcome: Group 2 - Number of Subjects With Absence of Radiolucency/Bone Loss
Description: Independent radiographic was performed on all required post-operative follow-up intervals and a detailed report was provided at the completion of the study. Each case was expected to have anteroposterio (A/P) and lateral radiographs obtained at all postoperative assessments. An independent review of the radiographs was assessed for progressive radiolucencies over time. Per the protocol, radiographic outcomes are defined as "An absence of subsidence of greater than or equal to 2 millimeters and an absence of both osteolysis and radiolucencies greater than or equal to 2 millimeters as determined by an independent radiographic reviewer."
Time Frame: 5 year
Population: Only subjects with an evaluable endpoint at the applicable time frame interval were used to calculate the count of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Mobile Unilateral Group (Group 2) | LPS Flex Mobile Bilateral Group (Group 2)
Number analyzed (Participants) | 106 | 14
Participants | 90 | 14

3. Primary Outcome: Group 2 - Number of Subjects With Absence of Implant Revision
Description: Revision is defined as "No intended, actual, or planned removal of any component of the knee system."
Time Frame: 5 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Mobile Unilateral Group (Group 2) | LPS Flex Mobile Bilateral Group (Group 2)
Number analyzed (Participants) | 106 | 14
Participants | 103 | 14

4. Primary Outcome: Group 2 - Number of Subjects With Absence of Severe Knee-Related Complication
Description: All severe knee-related complications are determined by each study investigator. A severe adverse event is any undesirable experience associated with the use of the implant in a patient that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in persistent or significant disability or incapacity, or is a birth defect. A knee-related complication is an adverse event that has been classified by the investigator to have a relation to the knee.
Time Frame: 5 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Mobile Unilateral Group (Group 2) | LPS Flex Mobile Bilateral Group (Group 2)
Number analyzed (Participants) | 106 | 14
Participants | 105 | 14

5. Primary Outcome: Group 1 - Total Knee Society Score (KSS)
Description: as for outcome 1
Time Frame: 4 year, 5 year, 6 year, 8 year, and 10 year
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- LPS Flex Mobile (Group 1): Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee. Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in both knees. Subjects in this group received the LPS-Flex Fixed Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee and were enrolled in a previous Investigational Device Exemption study. Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee and were enrolled in a previous Investigational Device Exemption study.
Arm/Group | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
Number analyzed (Participants) | 77 | 69
score on a scale
  4 Year: number analyzed (Participants) | 10 | 9
  4 Year | 164.6 (32.9) | 184.4 (9.7)
  5 Year: number analyzed (Participants) | 10 | 12
  5 Year | 142.4 (32.2) | 142.6 (41.3)
  6 Year: number analyzed (Participants) | 40 | 38
  6 Year | 161.9 (28.1) | 169.3 (29.8)
  8 Year: number analyzed (Participants) | 60 | 54
  8 Year | 164.8 (31.0) | 172.0 (26.9)
  10 Year: number analyzed (Participants) | 53 | 41
  10 Year | 166.6 (25.5) | 170.8 (29.3)

6. Primary Outcome: Group 1 - Number of Subjects With Absence of Radiolucency/Bone Loss
Description: as for outcome 2
Time Frame: 10 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
Number analyzed (Participants) | 72 | 63
Participants | 65 | 62

7. Primary Outcome: Group 1 - Number of Subjects With Absence of Implant Revision
Description: Revision is defined as "No intended, actual, or planned removal of any component of the knee system."
Time Frame: 10 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
Number analyzed (Participants) | 77 | 69
Participants | 75 | 68

8. Primary Outcome: Group 1 - Number of Subjects With Absence of Severe Knee-Related Complication
Description: as for outcome 4
Time Frame: 10 year
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
Number analyzed (Participants) | 77 | 69
Participants | 75 | 67

ADVERSE EVENTS:
Time Frame: Group 2 (PAS Group) - Pre-op, 6 week, 6 month, 1 year, 2 year, 3 year, 4 year, and 5 year. Group 1 (Subjects in the previous IDE study who were eligible to participate in the PAS) - 4 year, 5 year, 6 year, 8 year, and 10 year
Groups:
- LPS Flex Mobile Unilateral (Group 2): Cases were enrolled into a short-term study (5 years) and consisted of cases eligible to receive the LPS-Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement. Subjects who were implanted with the study device in one knee were in the Unilateral Group.
- LPS Flex Mobile (Group 1): Subjects in this group received the LPS Flex Mobile Bearing Knee implanted by an orthopedic surgeon experienced in primary total knee replacement in one knee and were enrolled in a previous Investigational Device
Arm/Group | LPS Flex Mobile Unilateral (Group 2) | LPS Flex Mobile Bilateral (Group 2) | LPS Flex Fixed (Group 1) | LPS Flex Mobile (Group 1)
All-Cause Mortality (participants affected / at risk) | 7/106 | 0/14 | 1/77 | 1/69
Serious Adverse Events (participants affected / at risk) | 17/106 | 0/14 | 8/77 | 5/69
Other Adverse Events (participants affected / at risk) | 82/106 | 14/14 | 64/77 | 14/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LPS Flex Mobile Unilateral (Group 2) (N=106) | LPS Flex Mobile Bilateral (Group 2) (N=14) | LPS Flex Fixed (Group 1) (N=77) | LPS Flex Mobile (Group 1) (N=69)
COLON CANCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ILIAC CREST FUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR FUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CERVICAL FUSION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KNEE JOINT REPLACEMENT SURGERY (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CRAINIOTOMY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOTAL HIP JOINT REPLACEMENT (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
MYELOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATIENT TRIPPED AND FELL HYPERFLEXING HER KNEE AND HAD PAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEGENERATIVE JOINT DISEASE OF RIGHT HIP (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INCREASED SWELLING AND PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND DRAINAGE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST CANCER (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
POSTERIOR DISLOCATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BLADDER TUMORS (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUPERFICIAL HEMATOMA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE CANCER (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC BYPASS (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
KNEE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STROKE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIBIAL COMPONENT LOOSENING (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LPS Flex Mobile Unilateral (Group 2) (N=106) | LPS Flex Mobile Bilateral (Group 2) (N=14) | LPS Flex Fixed (Group 1) (N=77) | LPS Flex Mobile (Group 1) (N=69)
ACUTE BLOOD LOSS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ADHESIVE CAPSULITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALLERGIC REACTION (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALZHEIMERS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANEMIA (Vascular disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
ANKLE FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ANKLE PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANKLE TENDINITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
AORTIC ANEURYSM VALVE REPLACEMENT (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ARTHRALGIA SHOULDER (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BACK INJURY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 3 (6) | 3 (3)
BENIGN MOLE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BICEP TEAR (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BICEP TENDON STRAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLADDER INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BLISTERS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BRONCHITITS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BURNING IN LEGS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BURSITIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4) | 0 (0) | 2 (2) | 0 (0)
BUTTOCKS BRUISE FROM FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
BUTTOCKS PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CALF PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CALF STIFFNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARCINOMA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARPAL TUNNEL SYNDROME (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 0 (0) | 2 (3)
CARPOMETACARPAL ARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CATARACT SURGERY (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 2 (3) | 4 (5) | 0 (0) | 0 (0)
CHEST PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHOLECYSTECTOMY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHONDROMALACIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CLL (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONGESTIVE HEART FAILURE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CONTACT DERMATITIS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
CREPITATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DEEP VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
DEGENERATIVE DISC DISEASE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DEGENERATIVE JOINT DISEASE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
DELAY WOUND HEALING (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
DIMINSHED SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 9 (9) | 1 (1)
DISC BULGE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISLOCATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DISTAL RADIUS FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DROP FOOT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN ON KNEE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELBOW PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ELEVATED BLOOD GLUCOSE (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ETIOLOGY (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FACIAL BLEEDING (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAILED TOTAL HIP ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE FROM FALL (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEVER (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FIBROMYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FLEXION CONTRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FLUID IN KNEE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
FOOT INJURY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
FOOT PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
GAIT ANOMOLY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRIC ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROCNEMIUS RUPTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HAND ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
HAND NUMBNESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAND OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAND PAIN FROM FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAND PARESTHESIAS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HAND TENDON RELEASE (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
HEMATOMA (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HERNIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE FROM FALL (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HIP OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
HIP PAIN (Musculoskeletal and connective tissue disorders) | 8 (9) | 2 (2) | 1 (1) | 2 (4)
HIP TROCHANTERIC BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOGLYCEMIA (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
INCREASED TROPONIN (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
INSTABILITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2)
KIDNEY CANCER (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
KNEE ANKYLOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KNEE BUCKLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KNEE CLICKING (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
KNEE EFFUSION (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 3 (3) | 0 (0)
KNEE INFLAMMATION (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
KNEE OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 12 (12) | 2 (2) | 3 (4) | 4 (5)
KNEE PAIN (Musculoskeletal and connective tissue disorders) | 39 (54) | 7 (11) | 15 (18) | 12 (12)
KNEE PAIN FROM FALL (Injury, poisoning and procedural complications) | 7 (7) | 0 (0) | 6 (6) | 7 (7)
KNEE SCAR TISSUE (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
KNEE STIFFNESS (Musculoskeletal and connective tissue disorders) | 14 (15) | 1 (1) | 1 (1) | 0 (0)
KNEE STRESS FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
KNEE SUBLUXATION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
KNEE SWELLING (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
KNEE TENDONITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
L-4 FRACTURE FROM FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LAXITY SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEG EDEMA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LEG PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LENS BROKE FROM CATARACTS (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEUKOCYTOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOW H AND H IN AM HGL 8.3 H T 24.8 (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOW HEMOGLOBIN (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
LOW OXYGEN LEVELS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUMBAR PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LUPUS FLARE (Immune system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
MASTECTOMY (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MENISCUS TEAR (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
METATORSAL DISPLACEMENT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEUROPATHY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NUCLEUS PULPOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOLYTIC CHANGES OF TIBIAL PLATEAU (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOPENIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAIN FROM FALL (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
PATELLA CLUNK (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PATELLA FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERONEAL NERVE PALSY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PINCHED NERVE IN ARM AND NECK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PINCHED NERVE SHOULDER (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLANTAR FASCITIS (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PROSTATE CARCINOMA (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
PULMONARY EMBOLISM (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RADIOLUCENCY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
REFLUX (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RENAL INSUFFICIENCY (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RIB FRACTURE FROM FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ROTATOR CUFF SURGERY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ROTATOR CUFF TEAR (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
SCIATICA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SHORTNESS OF BREATH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SHOULDER ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SHOULDER INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 2 (2) | 3 (3)
SHOULDER STITCHES AFTER FALL (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SI JOINT PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
SIATICA PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SKIN INFECTION ON INCISION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SNAKE BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SPINAL LSP (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
SPINE ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPINE NERVE ROOT IMPINGEMENTS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SYNOVITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TENDINITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
THIGH PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
THYROID NODULE (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TIBIAL CYSTS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TORN MENISCUS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOTAL HIP ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOTAL KNEE ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2) | 0 (0) | 0 (0)
TOTAL SHOULDER ARTHROPLASTY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRAUMATIC BRAIN INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRIGGER FINGER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TUMOR EXCISION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ULCER (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VARISCOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VASCULITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VERTEBRAL FRACTURE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WEAKNESS IN FOOT (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WOUND DRAINAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
WRIST ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WRIST FRACTURE (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
WRIST MASS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WRIST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
YELLOW DRAINAGE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-06): https://cdn.clinicaltrials.gov/large-docs/95/NCT00854295/Prot_SAP_000.pdf